CLINICAL TRIAL: NCT00422305
Title: Assessment of Lung Structure and Function of Infants Born Prematurely
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Robert Tepper, Robert Tepper, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 0603-15
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Premature Birth; Bronchopulmonary Dysplasia; Asthma
Keywords: Infant, Premature; Bronchopulmonary dysplasia; asthma
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1-Healthy Infants: Group 1: The investigators will recruit 80 healthy infants born at > 37 weeks gestation, and between 2 and 36 months of age. Infants will be excluded for any of the following reasons:
  1. Congenital cardio-respiratory disease
  2. Hospitalization for respiratory illness
  3. Treatment with asthma medications
  4. Small for gestational age at birth
- 2-Healthy Infants computerized Tomography: Group 2: The investigators recruited 4 infants born at > 37 weeks gestation and they were evaluated between 2 and 36 months of age when scheduled for high resolution computed tomography (HRCT) imaging for non-respiratory medical problems. Subjects were enrolled and HRCT of the chest were obtained. Infants were excluded for the following reasons:
  1. Congenital cardio-respiratory disease
  2. Hospitalization for respiratory illness
  3. Treatment with asthma medications
- 3-Premature Infants: Group 3: The investigators have recruited 45 infants born prematurely at 23-35 weeks gestation. Subjects were evaluated at corrected age at between 2 and 24 months. The subjects had no oxygen requirements, and were clinically stable outpatients when evaluated. Infants were excluded for any of the following reasons:
  1. Congenital cardio-respiratory disease
  2. Severe developmental delay

SUMMARY:
The purpose of this study is to evaluate the growth of the lung and how easily gas can be taken up by the lung in healthy infants born at full term without any breathing problems and infants born prematurely.

DETAILED DESCRIPTION:
SPECIFIC AIM #1:

Determine the relationship between parenchymal tissue and alveolar volume with normal lung growth early in life.

We hypothesize that during the first two years of life that parenchymal surface area and alveolar volume increase with somatic growth; however, the ratio of surface area to volume remains constant, while ventilation within the lung becomes more homogenous.

SPECIFIC AIM #2:

Determine the pulmonary sequelae of premature birth and assess the effectiveness of early treatment strategies upon the pulmonary sequelae.

We hypothesize that premature birth impedes growth and development of the lung parenchyma and the airways. In addition, initiating continuous positive airway pressure (CPAP) and a permissive ventilatory strategy in very premature infants at birth will improve lung growth and lung function compared to treatment with early surfactant and conventional ventilation.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* 37 weeks or greater gestational age
* Age 2 to 36 months

Group 2:

* 37 weeks or greater gestational age having a CT scan for non-respiratory issues.
* Age 2-36 months

Group 3:

* 23-35 weeks gestational age

Exclusion Criteria:

Group 1 and Group 2:

* Congenital cardio-respiratory disease
* Hospitalization for respiratory illness
* Treatment with asthma medications
* Small for gestational age at birth

Group 3:

* Congenital cardio-respiratory disease
* Severe developmental delay

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be selected from Infant Lung Disease Clinics at Riley Hospital, flyer in the community, and the neonatal intensive care unit (NICU) at Riley Hospial for Children, Indiana University and Methodist Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2007-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Testing | day of testing
  Forced expiratory Flows, Single-breath diffusion capacity and alveolar volume

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Tepper, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States